CLINICAL TRIAL: NCT07111234
Title: Examining the Role of Cooling Agents in Oral Nicotine Pouches
Brief Title: Studying Flavors and Cooling Agents in Oral Nicotine Pouches to Understand User Preferences
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Brittney Keller-Hamilton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: OSU-24236; NCI-2025-04693 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-07-29; First posted 2025-08-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Carbon Monoxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In a double-blind, randomized crossover design, N=30 adult daily cigarette smokers will sample 4 ONPs with varying flavor and synthetic coolant properties. Participants are blinded to their study product(s) and will not be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Chill (WS-3 only) (Experimental): Participants receive Chill-flavored nicotine pouch over 10 minutes and will complete questionnaires assessing measures of product appeal, sensory ratings and an oral tobacco purchase task.
  Interventions: Procedure: Carbon Monoxide Measurement; Drug: Nicotine Oral Pouch; Other: Questionnaire Administration
- Menthol (menthol only) (Experimental): Participants receive Menthol-flavored nicotine pouch over 10 minutes and will complete questionnaires assessing measures of product appeal, sensory ratings and an oral tobacco purchase task.
  Interventions: Procedure: Carbon Monoxide Measurement; Drug: Nicotine Oral Pouch; Other: Questionnaire Administration
- Peppermint (menthol+WS-3) (Experimental): Participants receive Peppermint-flavored nicotine pouch over 10 minutes and will complete questionnaires assessing measures of product appeal, sensory ratings and an oral tobacco purchase task.
  Interventions: Procedure: Carbon Monoxide Measurement; Drug: Nicotine Oral Pouch; Other: Questionnaire Administration
- Smooth (no menthol or WS-3) (Experimental): Participants receive Smooth-flavored nicotine pouch over 10 minutes and will complete questionnaires assessing measures of product appeal, sensory ratings and an oral tobacco purchase task.
  Interventions: Procedure: Carbon Monoxide Measurement; Drug: Nicotine Oral Pouch; Other: Questionnaire Administration
- Usual brand cigarette visit (Experimental): Participants smoke their usual brand cigarette over 5 minutes and will complete questionnaires assessing measures of product appeal, sensory ratings and a tobacco purchase task.
  Interventions: Procedure: Carbon Monoxide Measurement; Other: Questionnaire Administration; Drug: Smoke usual brand cigarette

INTERVENTIONS:
Procedure: Carbon Monoxide Measurement — Ancillary studies
  Other Names: Carbon Monoxide; CMONOX
Drug: Nicotine Oral Pouch — Sample randomly-ordered ONPs
  Other Names: ZYN
  Arms: Chill (WS-3 only); Menthol (menthol only); Peppermint (menthol+WS-3); Smooth (no menthol or WS-3)
Other: Questionnaire Administration — Ancillary studies
Drug: Smoke usual brand cigarette — Participant will smoke their usual brand of cigarette during 1 study visit for 5 minutes.
  Arms: Usual brand cigarette visit

SUMMARY:
This clinical trial studies how the flavors and synthetic coolant properties in oral nicotine pouches (ONPs) compare to one another and how these characteristics are perceived by users. ONPs are placed between the gum and lip, and the nicotine is absorbed in the mouth. They have a strong potential for harm reduction if smokers can switch to using them, and they are growing in popularity. One factor that could be contributing to the increase in popularity is the wide range of flavors, including mint or menthol. With recent flavor restriction policies that have gone into effect in certain areas of the United States, ONPs are now including synthetic cooling agents (WS-3) in place of the flavors. They provide a cooling sensation, but do not have a characterizing flavor, like mint or menthol, allowing them to be sold where flavor restriction policies are in place. Learning more about the flavors and cooling properties in ONPs and user preferences may help researchers guide future ONP regulation and understand how these characteristics may be used as a potential harm reduction or quit smoking tool.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the individual and joint effects of menthol flavors and WS-3 on appeal of ONPs.

II. Test the individual and joint effects of menthol flavors and WS-3 on self-reported relief of withdrawal and craving symptoms associated with use of ONPs.

II. Compare demand for ONPs that vary according to menthol flavors and WS-3.

OUTLINE: Participants are randomized to sample 4 ONPs in a 1 visit, 4-session, randomized cross-over study.

Participants sample four randomly-ordered ONPs with flavors consisting of WS-3 only, menthol only, menthol + WS-3, and no menthol or WS-3 over 10 minutes each, with washout periods of 10 minutes between each ONP use period.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Willing to complete study procedures, including abstaining from all tobacco, nicotine, and marijuana for 12 hours before clinic visits
* Ability to read and speak English
* Has smoked >= 100 cigarettes
* Smokes >= 5 cigarettes/day for past year

Exclusion Criteria:

* Use other tobacco products (including ONPs) more than 10 days per month
* Unstable or significant psychiatric conditions (past and stable conditions allowed)
* Pregnant, planning to become pregnant, or breastfeeding (will be verified with urine pregnancy test before each visit)
* History of cardiac event or distress within the past 3 months
* Currently attempting to quit all tobacco use

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Appeal ratings | 5, 15, and 30 minutes after initial product use. To be completed during the cigarette visit.
  The modified Cigarette Evaluation Questionnaire (mCEQ) will assess subjective appeal. The 11-item mCEQ includes five subscales: Satisfaction, Psychological Reward, Aversion, Enjoyment, and Craving Reduction. Individual items are rated from 1 (not at all) to 7 (extremely likely) and are averaged to create each subscale also ranging from 1 to 7. Higher values indicate greater levels of satisfaction, reward, aversion, enjoyment, and craving reduction.
Sensory ratings | 5, 15, and 30 minutes after initial product use. To be completed on the day of the study visit. The visit will last approximately 2.5 hours
  Sensory ratings will be evaluated with the general Labeled Magnitude Scale (gLMS), a 5-item self-report measure completed following ONP use. Scores range from 0 (no sensation) to 100 (strongest imaginable) with higher scores indicating a greater sensation intensity.
Withdrawal and Craving | 0, 5, 15, and 30 minutes after initial product use.To be completed on the day of the study visit. The visit will last approximately 2.5 hours
  Nicotine withdrawal and craving will be assessed using the Minnesota Nicotine Withdrawal Scale (MNWS). MNWS is the sum of 8 items rated on a 5-point scale from 0 (none) to 4 (severe) with scores ranging from 0 to 32; MNWS Craving is a single item with scores ranging from 0 to 4, higher scores indicate greater withdrawal/craving.
Demand indices | At the end of each ONP sampling session. To be completed on the day of the study visit. The visit will last approximately 2.5 hours
  After product use, participants will complete a purchase task to assess demand indices including demand elasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Brittney L Keller-Hamilton, PhD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu